CLINICAL TRIAL: NCT07122765
Title: Effect of Caloric Content And Timing of Meal On Postprandial Substrate Oxidation And Pulse Wave Analysis
Acronym: MetChrono
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NCR245996
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Feeding; Metabolism; Indirect Calorimetry; Blood Flow Velocity; Pulse Wave Analysis; Pulse Wave Velocity; Carbohydrate Metabolism; Fatty Acid Metabolism; Healthy Participants
Keywords: Feeding; postprandial; metabolism; pulse wave analysis

STUDY DESIGN:
Intervention Model Description: 3 arm randomized cross-over trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eucaloric Morning Mixed Meal Challenge (Active Comparator): Morning Mixed Meal Challenge (Liquid Shake), 25% of estimated daily caloric need
  Interventions: Other: Mixed Meal Feeding Challenge
- Eucaloric Evening Mixed Meal Challenge (Experimental): Evening Mixed Meal Challenge (Liquid Shake), 25% of estimated daily caloric need
  Interventions: Other: Mixed Meal Feeding Challenge
- Hypercaloric Morning Mixed Meal Challenge (Experimental): Morning Mixed Meal Challenge (Liquid Shake), 37.5% of estimated daily caloric need
  Interventions: Other: Mixed Meal Feeding Challenge

INTERVENTIONS:
Other: Mixed Meal Feeding Challenge — Liquid flavored Ensure Plus Shake of varying caloric content based on individual daily estimated caloric need

SUMMARY:
The overarching aim of this research is to study the effects of caloric content and timing of meals on measures of postprandial metabolism and cardiovascular response

1. Determine the effect of caloric content on measures of postprandial metabolic flexibility and pulse wave analysis to a mixed meal challenge.
2. Determine the effect of meal timing on measures of postprandial metabolic flexibility and pulse wave analysis to a mixed meal challenge.

Hypothesis: 1) that hypercaloric meals will result in significantly reduced indices of metabolic flexibility and pulse wave analysis as compared to eucaloric meals and 2) eucaloric meals consumed later in the day will result in significantly reduced metabolic flexibility and pulse wave analysis as compared to eucaloric meals consumed in the morning.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females between the ages of 18 and 45 years
* Low risk for medical complications as determined by physical activity readiness questionnaire (PARQ).
* Not currently taking antioxidant supplementation, non-steroidal anti-inflammatory drugs (NSAIDS) in a prescribed manner, antibiotics, steroids, or probiotics.
* Not currently taking any medications for management of cholesterol, diabetes, or body weight/obesity, or are undergoing transgender hormone therapy.
* Not currently pregnant
* No history of disordered eating, including anorexia nervosa, bulimia nervosa, binge eating disorder, or avoidant restrictive food intake disorder or screened as high risk for disordered eating via validated questionnaire.
* No history of gastrointestinal diseases, such as gastroesophageal reflux disease (GERD), irritable bowel syndrome, Celiac disease, Crohn's disease, or lactose intolerance.
* Considered low risk for food insecurity via the Hunger Vital Sign screener.
* Cannot have followed a ketogenic diet within the last three months or have been told to avoid a high-fat diet by a medical provider due to cardiovascular disease risk.

Exclusion Criteria:

* Are currently taking any antioxidant supplementation (daily multivitamin not included), prescribed non-steroidal anti-inflammatory drugs (NSAIDS), antibiotics, steroids, or probiotics.
* Are currently taking any medications for management of cholesterol, diabetes, or body weight/obesity, or are undergoing hormone therapy (oral contraceptives not included).
* Are unwilling or unable to comply with study procedures, at the discretion of the investigators.
* Pregnant women - A urine pregnancy test will be conducted prior to any testing procedures.
* A history of disordered eating, including anorexia nervosa, bulimia nervosa, binge eating disorder, or avoidant restrictive food intake disorder or deemed high-risk for disordered eating via questionnaire.
* A history of gastrointestinal diseases, such as gastroesophageal reflux disease (GERD), irritable bowel syndrome (IBS), Celiac disease, Crohn's disease, or lactose intolerance.
* Deemed high risk for food insecurity via the Hunger Vital Sign screener which is filled out electronically prior to enrollment.
* Have followed a ketogenic diet within the last three months or have been told to avoid a high-fat diet by a medical provider for risk of cardiovascular disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulse Wave Analysis | Baseline to 60 and 120 minutes postprandial
  Augmentation Index normalized to 75 beats per minute as index of pulse wave reflection
Postprandial Substrate Oxidation | Baseline to 120 minutes postprandial
  Respiratory Exchange Ratio

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington University School of Public Health, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data will be shared with researchers upon resonable request and data will be deposited on Open Science Framework
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: June 2026 upon completion of primary data collection and analysis of primary outcomes
Access Criteria: Researchers making reasonable requests for data access will be granted permission and access to primary data files. Researchers will be asked to submit a scientific question and rationale for data access along with a data analysis plan. Researchers will intiiate a Data Use Agreement with Principal Investigators.